CLINICAL TRIAL: NCT04214366
Title: Adenoid Cystic Carcinoma and Carbon Ion Only Irradiation
Acronym: ACCO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Klaus Herfarth, MD, Prof. Dr. Klaus Herfarth, Vice chair Dept. of Radiation Oncology, Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACCO
Record Dates: First submitted 2019-09-24; First posted 2020-01-02 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Adenoid Cystic Carcinoma
Keywords: carbon ion; heavy ion; salivary gland tumor; ACC; Radiation therapy
MeSH Terms: conditions — Carcinoma, Adenoid Cystic; Salivary Gland Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carbon Ion irradiation (Experimental): 22 x 3 Gy(RBE) Carbon Ions
  Interventions: Radiation: Carbon ion irradiation
- Bimodal Arm (Active Comparator): 25 x 2 Gy photon IMRT and 8 x 3 Gy(RBE) Carbon ion boost
  Interventions: Radiation: Bimodal irradiation

INTERVENTIONS:
Radiation: Carbon ion irradiation — 22 x 3 Gy(RBE) Carbon Ions
  Arms: Carbon Ion irradiation
Radiation: Bimodal irradiation — 25 x 2 Gy photon IMRT + 8 x 3 Gy(RBE) Carbon ion boost
  Arms: Bimodal Arm

SUMMARY:
Adenoid cystic tumors are rare tumors of the head and neck region. Despite their slow growth, re-irradiation is often necessary due to the high metastatic risk. Patients are usually irradiated with photons or, as here at the Heidelberg University Hospital, with a combination of carbon ions and photons. So far, there is no data from Europe available for the sole irradiation with carbon ions. The present ACCO (Adenoid Cystic Carcinoma and Carbon ion Only irradiation) study, a prospective, open-label, phase II, single-arm, investigator-initiated study, will therefore investigate the sole radiotherapy of carbon ions in this tumor entity. Irradiation is applied - significantly shorter than the combination therapy - in about 4 weeks (22 fractions); patients are followed up for further 5 years after the start of therapy. Carbon ions alone are expected to increase local tumor control rates from 60% to 70% after 5 years (primary objective criterion of this study). In order to reject the null hypothesis with a power of 80% and a significance level of 5%, 175 patients are included (including a drop-out rate of 15%). Secondary objective criteria are progression-free survival, overall survival, acute and late toxicity, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenoid cystic carcinoma in the head and neck area
* Indication for irradiation:
* non-operable or
* R1/R2 resected or
* perineural sheat invasion (Pn+) or
* pT3/pT4
* Informed consent
* KI > 60% or ECOG 0/1 (minimum: self-sufficiency, normal activity or work not possible)
* Age 18-80 years

Exclusion Criteria:

* rejection of the study by the patient
* Patient is not able to consent
* Stage IV (distant metastases), except lung metastases < 1cm
* lymph node involvement (clinical or pathological)
* Previous radiotherapy in the head and neck area
* Active medical implants for which there is no ion radiation authorization at the time of treatment (e.g., cardiac pacemaker, defibrillator, ...)
* Contraindication to MR imaging
* Simultaneous participation in another clinical study that could influence the outcome of this study or the other study
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2032-12-01 (Estimated)

PRIMARY OUTCOMES:
Freedom from loco-regional progression | at 5 years
  Freedom from loco-regional tumor progression according to MR imaging

SECONDARY OUTCOMES:
Progression-free survival | at 3 and 5 years
  Progression-free survival
Overall survival | at 3 and 5 years
  Overall survival
Acute toxicities | during and up to 6 weeks after radiotherapy
  Acute toxicities according to NCI CTC AE (Version 5.0) (rate of toxicity > 2 grade)
Late toxicities | up to 5 years
  Late toxicities according to NCI CTC AE (Version 5.0) (rate of toxicity > 2 grade)

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Herfarth, Prof. Dr., Principal Investigator — University Hospital Heidelberg
Locations (1):
- University of Heidelberg, Radiooncology, HIT, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lang K, Adeberg S, Harrabi S, Held T, Kieser M, Debus J, Herfarth K. Adenoid cystic Carcinoma and Carbon ion Only irradiation (ACCO): Study protocol for a prospective, open, randomized, two-armed, phase II study. BMC Cancer. 2021 Jul 15;21(1):812. doi: 10.1186/s12885-021-08473-5. PMID 34266402

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/66/NCT04214366/Prot_SAP_000.pdf